CLINICAL TRIAL: NCT02614989
Title: MRI Guided Focused Ultrasound for Tremor in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0556-15-RMB
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
Keywords: Tremor; Thalamotomy
MeSH Terms: conditions — Multiple Sclerosis; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI guided Focused Ultrasound treatment (Experimental): MRI guided focused ultrasound thalamotomy
  Patients will undergo unilateral thalmotomy using MRI guided Focused Ultrasound intervention for the treatment of the tremor
  Interventions: Procedure: MRI guided focused ultrasound thalamotomy

INTERVENTIONS:
Procedure: MRI guided focused ultrasound thalamotomy — MRI guided focused ultrasound thalamotomy

SUMMARY:
This project goal is to explore the option of (MRgFUS) as a treatment for tremor in MS patients with disabling refractory tremor.

DETAILED DESCRIPTION:
This study is designed as a prospective, single site, single arm, nonrandomized study. Assessments will be made before and after MRgFUS for clinical symptom relief, quality of life (QoL) improvements, and safety of MRgFUS in the treatment of multiple sclerosis patients with severe medication refractory tremor.

This study will be performed on the 3T MR scanners. The ExAblate system is a medical device that involves a focused ultrasound system and an MRI scanner. During MRgFUS a pulse of focused ultrasound energy, or sonication,are delivered to the targeted tissue. In this particular study the targeted tissue is a unilateral thermal lesion created in the ventralis intermedius nucleus of the thalamus.

The treatment begins with a series of standard diagnostic MR images to identify the location and shape of tumor to be treated. The computer uses the physician's designation of the target volume to plan the best way to cover the target volume with small spots called "sonications". These treatment spots are cylinder shaped. Their size depends on sonication power and duration. During the treatment, a specific MR scan, which can be processed to identify changes in tissue temperature, provides a thermal map of the treatment volume to confirm the therapeutic effect. The thermal map is used to monitor the treatment in progress, and confirm that the ablation is proceeding according to plan, thus closing the therapy loop.

MRgFUS uses a transcranial operated helmet-shaped transducer positioned above the subject head. The transcranial system includes means to immobilize the subject head, cool the interface water, and software for CT analysis and phase correction computation.

MRgFUS transcranial system to relieve tremor in multiple sclerosis patients is being investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 years and older
* Patients who are able and willing to give informed consent and able to attend all study visits
* Patients with a diagnosis of Multiple sclerosis (MS) as confirmed from clinical history and examination by a neurologist.
* The patient must have disabling tremor from MS as indicated by a score of at least 2 on the Tremor Rating Scale (TRS) baseline global assessments by the examiner and the patient. Or Disabling is defined as significant impairment of the normal functions of daily life as indicated by a score of at least 5 on the Clinical Global Impression (CGI)-Severity scale.or ETRS
* The MS patient must have disabling and medically refractory unilateral or bilateral upper extremity tremor. Patients with associated ipsilateral lower extremity tremor are not excluded.
* The patient must have a history of an unsatisfactory response to medical management. Any patient will need to have tried and failed at least one drug. Alternatively, a patient may also qualify if tremor-suppressing medications are contraindicated due to a coexisting medical condition or drug allergy.
* Patients should be on a stable dose of medications for 30 days prior to study entry

Exclusion Criteria:

* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Significant claustrophobia
* Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment
* Subjects with unstable cardiac status
* Severe hypertension
* Current medical condition resulting in abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within two weeks of focused ultrasound procedure or drugs known to increase risk or hemorrhage
* History of intracranial hemorrhage
* History of multiple strokes, or a stroke within past 6 months
* Subjects with a history of seizures within the past year
* Subjects with brain tumors
* Are participating or have participated in another clinical trial in the last 30 days
* More than mild non-tremor cerebellar dysfunction (ataxia, dysmetria, dysdiadokokinesia).
* Cognitive dysfunction as evidenced by a score of less than ??? on the ???

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Device or procedure related adverse events reported | 3 months
  Safety of the MRI guided focused Ultrasound treatment will be determined by an evaluation of the incidence and severity of device and procedure related complications from the first / treatment day visit through the 3-Months post-treatment time point. All AEs will be reported.

SECONDARY OUTCOMES:
Tremor rating scale | 1 month
  Tremor Rating Scale